CLINICAL TRIAL: NCT01402310
Title: Bishop Score, Cervical Length and Multiple Proteins in Cervicovaginal Fluid at 40 Weeks to Predict Onset of Labor
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BS_CL_40wk
Record Dates: First submitted 2011-03-17; First posted 2011-07-26 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Prolonged Labor
Keywords: Onset of labor; Bishop score; Cervical length; Multiple proteins; Cervicovaginal fluid
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cervicovaginal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women attending antenatal clinic: Women attending antenatal clinic were consecutively enrolled at between 39+6 and 40+1 weeks of gestation.
  Interventions: Other: Ultrasound and digital cervical examination

INTERVENTIONS:
Other: Ultrasound and digital cervical examination — Cervical length by transvaginal ultrasound Bishop score by digital examination Take cervicovaginal samples

SUMMARY:
The purpose of this study is to compare Bishop score, sonographic cervical length and multiple proteins in cervicovaginal fluid at 40 weeks gestation to predict time to spontaneous labor and mode of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women between 39+6 and 40+1 weeks of gestation
* singleton pregnancy
* viable fetus with vertex presentation
* intact amniotic membranes
* no pregnancy complications
* absence of labor
* no history of previous uterine surgery
* planned vaginal delivery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Single tertiary hospital
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2008-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Onset of labor/delivery ≤10days | Baseline

SECONDARY OUTCOMES:
Cesarean delivery in labor | Baseline
  1. Time to onset of spontaneous labor
  2. Postterm delivery (≥40 + 11 weeks of pregnancy)
  3. The rate of cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Hoon Park, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Obstetrics and Gynecology Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea